CLINICAL TRIAL: NCT01557348
Title: A Global Multi-centre Observational Study in RA Patients Who Are Non Responders or Intolerant to a Single TNF Inhibitor.
Brief Title: An Observational Study of MabThera/Rituxan (Rituximab) and Alternative TNF-Inhibitors in Patients With Rheumatoid Arthritis and an Inadequate Response to a Single Previous TNF-Inhibitor
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MA22401
Record Dates: First submitted 2012-03-13; First posted 2012-03-19 (Estimated); Results first posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Rituximab: Eligible participants will receive rituximab as second biologic therapy in routine clinical practice and were observed for 12 months from the start of the second biologic therapy.
- Alternative TNFi: Eligible participants will receive alternative TNFi treatment as second biologic therapy in routine clinical practice and were observed for 12 months from the start of the second biologic therapy.

SUMMARY:
This multicenter, prospective, observational study will assess the efficacy of MabThera/Rituxan (rituximab) and alternative TNF-inhibitors in patients with rheumatoid arthritis who are non-responders or intolerant to a single previous TNF-inhibitor. Data will be collected from each patient from the time of change in biologic therapy for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Patients with rheumatoid arthritis (RA) who have not responded or have been intolerant to a single TNF-inhibitor therapy
* Initiated on treatment with MabThera/Rituxan or an alternative TNF-inhibitor therapy, in accordance with the relevant Summary of Product Characteristics

Exclusion Criteria:

* Patients whose second biologic therapy is given as part of a clinical trial studying RA treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients who are non-responders or intolerant to a single TNF-inhibitor
Sampling Method: Probability Sample
Enrollment: 1239 (Actual)
Dates: Start 2009-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (182):
- Canada (14):
  - Winnipeg, Manitoba
  - Saint John, New Brunswick
  - Brampton, Ontario
  - Burlington, Ontario
  - Hamilton, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - St. Catharines, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Rimouski, Quebec
  - Saskatoon, Saskatchewan
- Colombia (3):
  - Barranquilla
  - Bogotá
  - Cali
- France (73):
  - Abbeville
  - Aix-les-Bains
  - Amiens
  - Argenteuil
  - Bayonne
  - Belfort
  - Besançon
  - Bonneville
  - Bordeaux
  - Boulogne-Billancourt
  - Brest
  - Bruges
  - Bry-sur-Marne
  - Caen
  - Cahors
  - Cambrai
  - Cannes
  - Carcassonne
  - Carhaix-Plouguer
  - Chambray-lès-Tours
  - Clermont-Ferrand
  - Colmar
  - Corbeil-Essonnes
  - Draguignan
  - Échirolles
  - Évreux
  - Issy-les-Moulineaux
  - La Roche-sur-Yon
  - La Source
  - Laon
  - Laval
  - Le Coudray
  - Le Kremlin-Bicêtre
  - Le Mans
  - Libourne
  - Liévin
  - Lille
  - Limoges
  - Lomme
  - Lorient
  - Lyon
  - Maisons-Laffitte
  - Mantes-la-Jolie
  - Marseille
  - Mennecy
  - Metz
  - Montauban
  - Montivilliers
  - Montpellier
  - Mulhouse
  - Nantes
  - Nevers
  - Nice
  - Pachuca
  - Paris
  - Perpignan
  - Pierre-Bénite
  - Reims
  - Rennes
  - Rodez
  - Roubaix
  - Saint-Aubin-lès-Elbeuf
  - Saint-Brieuc
  - Saint-Priest-en-Jarez
  - Toulon
  - Toulouse
  - Tours
  - Valence
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Vannes
  - Villeneuve-sur-Lot
  - Vincennes
- Germany (14):
  - Aachen
  - Bremen
  - Cologne
  - Cuxhaven
  - Erlangen
  - Frankenberg
  - Frankfurt
  - Gräfelfing
  - Halle
  - Hanover
  - Münster
  - Neuss
  - Rostock
  - Villingen-Schwenningen
- Greece (2):
  - Athens
  - Larissa
- Italy (20):
  - Coppito, Abruzzo
  - Bari, Apulia
  - San Cesario di Lecce, Apulia
  - Potenza, Basilicate
  - Napoli, Campania
  - Telese Terme, Campania
  - Ferrara, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Milan, Lombardy
  - Gazzi, Sicily
  - Palermo, Sicily
  - Ancona, The Marches
  - Iesi, The Marches
  - Florence, Tuscany
  - Pisa, Tuscany
  - Prato, Tuscany
  - Siena, Tuscany
  - Padua, Veneto
  - Verona, Veneto
- Mexico (4):
  - Chihuahua City
  - Mexicali
  - Mexico City
  - Poza Rica Chacas
- Monaco, Monaco
- Ålesund, Norway
- Portugal (4):
  - Amadora
  - Guimarães
  - Lisbon
  - Porto
- Spain (10):
  - Córdoba, Cordoba
  - Granada, Granada
  - León, Leon
  - Lugo, Lugo
  - Madrid, Madrid
  - El Palmar, Murcia
  - Lorca, Murcia
  - Salamanca, Salamanca
  - Seville, Sevilla
  - Torrevieja
- United Kingdom (36):
  - Abergavenny
  - Aylesbury
  - Blackburn
  - Cambridge
  - Cannock
  - Cardiff
  - Cheltenham
  - Chertsey
  - Cosham
  - Derby
  - Durham
  - Exeter
  - Glasgow
  - Harrogate
  - Inverness
  - Lancaster
  - Leeds
  - Lincoln
  - Liverpool
  - London
  - Manchester
  - Metropolitan Borough of Wirral
  - Poole
  - Salford
  - Solihull
  - Southport
  - St Helens
  - Stockport
  - Sunderland
  - Sutton in Ashfield
  - Torquay
  - Truro
  - Warrington
  - Wolverhampton
  - Worthing
  - Wrightington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study was conducted in 11 countries from 02 June 2009 to 19 March 2012.
Pre-assignment Details: Of 1239 enrolled participants, 9 had no information on second biologic treatment/reasons for discontinuing prior tumor necrosis factor inhibitor (TNFi), 1111 had one previous TNFi,119 had more than one previous TNFi. Of 1111 participants, 728 were considered for primary effectiveness analysis (405 in Rituximab arm and 323 in Alternative TNFi arm).
Groups:
- Rituximab: Eligible participants received rituximab as second biologic therapy in routine clinical practice and were observed for 12 months from the start of the second biologic therapy.
- Alternative TNFi: Eligible participants received alternative TNFi treatment as second biologic therapy in routine clinical practice and were observed for 12 months from the start of the second biologic therapy.
Period: Overall Study
Arm/Group | Rituximab | Alternative TNFi
Started | 604 | 507
Safety Population | 604 | 507
Completed | 524 | 417
Not Completed | 80 | 90
Not completed — Adverse Event | 6 | 16
Not completed — Infusion reaction event | 5 | 5
Not completed — Death | 7 | 4
Not completed — Insufficient Therapeutic Response | 13 | 28
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 26 | 22
Not completed — Administrative | 18 | 11

BASELINE CHARACTERISTICS:
Population: The primary effectiveness population included all participants who received at least one dose of a second biologic therapy at baseline (day of change in biologic therapy [<=Day 1]), had only one previous biologic therapy, and contributed for 24-week disease activity score 28 (DAS28)-erythrocyte sedimentation rate (ESR) for primary analysis.
Groups:
- Alternative TNFi: Eligible participants received alternative TNFi as second biologic therapy in routine clinical practice and were observed for 12 months from the start of the second biologic therapy.
- Total: Total of all reporting groups
Arm/Group | Rituximab | Alternative TNFi | Total
Number analyzed (Participants) | 405 | 323 | 728
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (12.61) | 54.7 (13.26) | 55.7 (12.93)
Gender [Count of Participants; unit: Participants]
  Female | 310 | 259 | 569
  Male | 95 | 64 | 159

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Change From Baseline in Disease Activity Score (3 Variables)-Erythrocyte Sedimentation Rate at Month 6
Description: The DAS28-3 (ESR) is a measure of disease activity in rheumatoid arthritis. It is calculated from the number of swollen joint count (SJC) and tender joint count (TJC) using the 28 joints count, and ESR (millimeters per hour [mm/hr]). Total score ranges from 0 to 9.4, where higher score indicated more disease activity. Decrease in score indicated improvement in disease activity.
Time Frame: Baseline (Day of change in biologic therapy [<=Day 1]) and Month 6
Population: The primary effectiveness population included all participants who received at least one dose of a second biologic therapy at Baseline, had only one previous biologic therapy, and contributed to 24-week DAS28-ESR primary endpoint analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 405 | 323
scores on a scale | -1.5 (0.22) | -1.1 (0.23)
Statistical Analysis 1: Comparison: Rituximab vs Alternative TNFi; Test type: Superiority or Other; p = 0.0068, ANCOVA — LsMean and p-value are based on an ANCOVA model adjusted for significant factors leading to selection of new biologic therapy and unbalanced baseline covariates

2. Secondary Outcome: Least Squares Mean Change From Baseline in Disease Activity Score (3 Variables)-Erythrocyte Sedimentation Rate at Month12
Description: as for outcome 1
Time Frame: Baseline (Day of change in biologic therapy [<=Day 1]) and Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 332 | 266
scores on a scale | -1.5 (0.27) | -1.2 (0.29)
Statistical Analysis 1: Comparison: Rituximab vs Alternative TNFi; Test type: Superiority or Other; p = 0.0588, ANCOVA — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Least Squares Mean Change From Baseline in TJC at Months 6 and 12
Description: The TJC is the most specific clinical method to quantify abnormalities in participants with rheumatoid arthritis (RA). A total of 28 joints were assessed for tenderness. Decrease in score indicated an improvement in disease activity.
Time Frame: Baseline, Month 6, and Month 12
Population: The primary effectiveness population included all participants who received at least one dose of a second biologic therapy at Baseline, had only one previous biologic therapy, and contributed to 24-week DAS28-ESR primary endpoint analysis. Participants with available data at specified time points were analyzed and are denoted as 'n'.
Measure: Least Squares Mean (Standard Error); unit: tender joints
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 338 | 255
tender joints
  Month 6 (n= 338, 255) | -5.7 (1.20) | -4.5 (1.24)
  Month 12 (n= 281, 216) | -4.7 (1.29) | -3.7 (1.36)
Statistical Analysis 1: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in TJC at Month 6; Test type: Superiority or Other; p = 0.1126, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in TJC at Month 12; Test type: Superiority or Other; p = 0.2342, ANCOVA — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Least Squares Mean Change From Baseline in SJC at Months 6 and 12
Description: The SJC is the most specific clinical method to quantify abnormalities in participants with RA. A total of 28 joints were assessed for swelling. Decrease in the score indicated improvement in disease activity.
Time Frame: Baseline, Month 6, and Month 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: swollen joints
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 339 | 256
swollen joints
  Month 6 (n= 339, 256) | -3.3 (0.93) | -2.8 (0.97)
  Month 12 (n= 283, 215) | -2.7 (0.99) | -2.4 (1.04)
Statistical Analysis 1: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in SJC at Month 6; Test type: Superiority or Other; p = 0.4168, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in SJC at Month 12; Test type: Superiority or Other; p = 0.5867, ANCOVA — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Least Squares Mean Change From Baseline in C-reactive Protein at Months 6 and 12
Description: C-reactive protein (CRP) is an inflammation marker. Normal range is from 0-10 milligram/Liter. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement in disease activity.
Time Frame: Baseline, Month 6, and Month 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: milligram/Liter
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 278 | 227
milligram/Liter
  Month 6 (n= 278, 227) | -29.1 (7.95) | -29.9 (8.43)
  Month 12 (n=251, 199) | -11.6 (8.47) | -15.3 (8.91)
Statistical Analysis 1: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in CRP at Month 6; Test type: Superiority or Other; p = 0.8758, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in CRP at Month 12; Test type: Superiority or Other; p = 0.4849, ANCOVA — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Least Squares Mean Change From Baseline in ESR at Months 6 and 12
Description: The ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells sediment in a period of one hour. Normal range is 0-30 mm/hr. A reduction in the level of ESR is considered as an improvement in disease activity.
Time Frame: Baseline, Month 6, and Month 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm/hr
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 343 | 250
mm/hr
  Month 6 (n= 343, 250) | -13.2 (3.91) | -7.0 (4.22)
  Month 12 (n=297, 215) | -11.6 (4.58) | -8.6 (4.90)
Statistical Analysis 1: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in ESR at Month 6; Test type: Superiority or Other; p = 0.0086, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in ESR at Month 12; Test type: Superiority or Other; p = 0.2918, ANCOVA — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Least Squares Mean Change From Baseline in Physician Global Assessment of Disease at Months 6 and 12
Description: Physician global assessment of disease was measured on a 0 to 100 millimeter (mm) visual analog scale (VAS), with 0 mm = no disease activity and 100 mm = highest possible disease activity. Higher scores indicate worsening of disease.
Time Frame: Baseline, Month 6, and Month 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 203 | 169
mm
  Month 6 (n= 203, 169) | -21.0 (6.13) | -14.8 (6.65)
  Month 12 (n= 169, 144) | -21.8 (6.69) | -14.3 (7.30)
Statistical Analysis 1: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in Physician Global Assessment of Disease at Month 6; Test type: Superiority or Other; p = 0.0764, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in Physician Global Assessment of Disease at Month 12; Test type: Superiority or Other; p = 0.0587, ANCOVA — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Least Squares Mean Change From Baseline in Patient Global Assessment of Disease at Months 6 and 12
Description: Patient Global Assessment of Disease was measured on a 0 to 100 mm VAS, with 0 mm = no disease activity and 100 mm = highest possible disease activity. Higher scores indicate worsening of disease.
Time Frame: Baseline, Month 6, and Month 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 288 | 219
mm
  Month 6 (n= 288, 219) | -17.0 (5.48) | -10.2 (5.77)
  Month 12 (n= 242, 189) | -19.7 (5.85) | -17.1 (6.24)
Statistical Analysis 1: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in Patient Global Assessment of Disease at Month 6; Test type: Superiority or Other; p = 0.0443, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in Patient Global Assessment of Disease at Month 12; Test type: Superiority or Other; p = 0.4802, ANCOVA — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Least Squares Mean Change From Baseline in Participant's VAS Pain Score at Months 6 and 12
Description: Participants were asked to assess their pain intensity (severity of pain) on a 100-millimeter (mm) VAS with the left edge (0 mm) defined as "no pain" and the right edge (100 mm) defined as "severest pain". Higher scores indicate worsening of disease.
Time Frame: Baseline, Month 6, and Month 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 236 | 197
mm
  Month 6 (n= 236, 197) | -15.7 (6.48) | -10.8 (7.02)
  Month 12 (n=194, 171) | -19.0 (6.58) | -10.0 (7.10)
Statistical Analysis 1: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in Participant's Visual Analogue Scale Pain Score at Months 6; Test type: Superiority or Other; p = 0.2026, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in Participant's Visual Analogue Scale Pain Score at Months 12; Test type: Superiority or Other; p = 0.0295, ANCOVA — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Least Squares Mean Change From Baseline in Health Assessment Questionnaire-Disability Index at Months 6 and 12
Description: Health Assessment Questionnaire-Disability Index (HAQ-DI) is participant reported assessment of ability to perform tasks in 8 categories of daily living activities as dress/groom, arise, eat, walk, reach, grip, hygiene, and common activities over past week. Each item was scored on a 4-point scale from 0 to 3, where 0=no difficulty, 1=some difficulty, 2=much difficulty, and 3=unable to do. Overall score was computed as the sum of domain scores divided by the number of domains answered. Total possible score range was 0-3, where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Month 6, and Month 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 164 | 131
scores on a scale
  Month 6 (n= 164, 131) | -0.6 (0.18) | -0.5 (0.19)
  Month 12 (n=142, 112) | -0.3 (0.20) | -0.2 (0.22)
Statistical Analysis 1: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in HAQ-DI at Month 6; Test type: Superiority or Other; p = 0.3370, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in HAQ-DI at Month 12; Test type: Superiority or Other; p = 0.1515, ANCOVA — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Least Squares Mean Change From Baseline in Duration of Morning Stiffness at Months 6 and 12
Description: Duration of morning stiffness is defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes. Participants with available data at the time of assessment were included in the analysis.
Time Frame: Baseline, Month 6, and Month 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 233 | 180
minutes
  Month 6 (n= 233, 180) | -19.0 (25.38) | -4.3 (27.37)
  Month 12 (n=206, 156) | -16.7 (25.81) | -1.4 (28.19)
Statistical Analysis 1: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in duration of morning stiffness at month 6; Test type: Superiority or Other; p = 0.3253, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Rituximab vs Alternative TNFi; Comparison of least squares mean change from Baseline in duration of morning stiffness at month 12; Test type: Superiority or Other; p = 0.3535, ANCOVA — [p-value comment as in outcome 1, analysis 1]

12. Secondary Outcome: Percentage of Participants Who Remained on Their Second Biologic Therapy at Months 6 and 12 After Start of Second Biologic Therapy
Description: Percentage of participants who remained on their second biologic therapy at 6 and 12 months after start of second biologic therapy were reported.
Time Frame: Month 6 and Month 12
Population: Safety analysis population included all enrolled participants with only one previous TNFi whose second biologic therapy (i.e,Treatment Group) and reason for changing biologic therapy was known.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 604 | 507
Percentage of participants | NA — The data recorded on the eCRF was insufficient to determine this outcome measure. The data recorded on the eCRF was insufficient for us to be able to determine this measure. | NA — The data recorded on the eCRF was insufficient to determine this outcome measure.

13. Secondary Outcome: Reasons for Stopping the Second Biologic Therapy and Subsequent Therapy Choice
Time Frame: Up to 12 months
Population: Safety analysis population included all enrolled participants with only one previous TNFi whose second biologic therapy (ie,Treatment Group) and reason for changing biologic therapy was known.
Measure: Number; unit: Number of participants
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 604 | 507
Number of participants | NA — Data was not actually collected as per the eCRF | NA — Data was not actually collected as per the eCRF

14. Secondary Outcome: Number of Participants With Any Adverse Events, Any Serious Adverse Event, Adverse Events Leading to Withdrawal, and Death
Description: An Adverse event is defined as any unfavorable and unintended medical occurrence/sign (including an abnormal laboratory finding), symptom or disease in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A serious adverse event is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: Up to 12 Months
Population: Safety analysis population included all enrolled participants with only one previous TNFi whose second biologic therapy and reason for changing biologic therapy was known.
Measure: Number; unit: participants
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 604 | 507
participants
  Any AE | 291 | 241
  Any SAE | 82 | 56
  AE leading to withdrawal | 17 | 39
  Death | 7 | 4

15. Secondary Outcome: Number of Participants With Reasons for Discontinuation of the First TNFi Therapy
Description: The reasons for discontinuation of first TNFi therapy included inefficacy, intolerance and other reasons. The other reasons included complete remission and participants' non-compliance.
Time Frame: Day 1 (Study entry visit)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 405 | 323
participants
  Inefficacy | 311 | 236
  Intolerance | 89 | 79
  Other reasons | 5 | 8

16. Secondary Outcome: Number of Participants With Previous TNFi Therapy
Description: The previous TNFi therapy included adalimumab, etanercept, infliximab, and others (certolizumab, and golimumab). Number of participants with previous TNFi therapy history was reported.
Time Frame: Day 1 (Study entry visit)
Population: The primary effectiveness population included all participants who received at least one dose of a second biologic therapy at baseline, had only one previous biologic therapy, and contributed to 24-week DAS28-ESR primary endpoint analysis. Participants with available data at specified time points are denoted as 'n'.
Measure: Number; unit: participants
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 405 | 323
participants
  Adalimumab (Humira) | 131 | 116
  Etanercept (Enbrel) | 176 | 162
  Infliximab (Remicade) | 95 | 42
  Certolizumab pegol (Cimzia) | 3 | 0
  Golimumab (Simponi) | 0 | 3

17. Secondary Outcome: Number of Participants With Previous Non-biologic Disease-modifying Anti-rheumatic Drugs Therapy
Description: The previous disease-modifying anti-rheumatic drugs therapy included auranofin, aurothioglucose, aurotioprol, azathioprine, chloroquine, ciclosporin, gold, hydroxychloroquine, infliximab, leflunomide, methotrexate, methotrexate sodium, minocycline, penicillamine, sodium aurothiomalate, sodium aurotiosulfate, sulfasalazine, and tiopronin. Number of participants with previous disease-modifying anti-rheumatic drugs therapy was reported.
Time Frame: Day 1 (Study entry visit)
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 405 | 323
participants
  Auranofin | 5 | 6
  Aurothioglucose | 0 | 1
  Aurotioprol | 4 | 4
  Azathioprine | 20 | 9
  Chloroquine | 27 | 11
  Ciclosporin | 25 | 27
  Gold | 27 | 20
  Hydroxychloroquine | 96 | 99
  Infliximab | 1 | 0
  Leflunomide | 144 | 126
  Methotrexate | 199 | 180
  Methotrexate sodium | 3 | 1
  Minocycline | 0 | 3
  Penicillamine | 7 | 5
  Sodium aurothiomalate | 17 | 4
  Sodium aurotiosulfate | 0 | 1
  Sulfasalazine | 107 | 86
  Tiopronin | 0 | 1

18. Secondary Outcome: Factors Related to Selection of Second Biologic Therapy Following an Insufficient Response or Intolerance to a Single Previous TNFi
Description: The factors included participant characteristics and the reasons that led to the selection of second biologic therapy following an insufficient response or intolerance to a single previous TNFi. The participant characteristics included participant's option for treatment and option for follow-up. The other reasons included RA disease (rheumatoid factor [RF] and cyclic citrullinated peptide [CCP] status), primary failure, and new treatment characteristics (rapidity of action, route of administration, frequency of administration, low infectious risk, and no lymphoma risk). Participants were included in more than one of these factors.
Time Frame: Baseline
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Rituximab | Alternative TNFi
Number analyzed (Participants) | 604 | 507
participants
  RA Disease (RF and CCP Status) | 344 | 216
  Primary failure | 256 | 135
  Rapidity of action | 82 | 203
  Route of administration | 123 | 289
  Frequency of administration | 303 | 174
  Low infectious risk | 172 | 62
  No lymphoma risk | 120 | 17
  Participant's option for treatment | 272 | 278
  Participant's option for follow-up | 91 | 89

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: All serious adverse events (SAEs) and non-serious adverse events (AEs) were reported for the safety population which included all participants who received a second biologic therapy at baseline and had one and only one previous biologic therapy.
Arm/Group | Rituximab | Alternative TNFi
Serious Adverse Events (participants affected / at risk) | 82/604 | 56/507
Other Adverse Events (participants affected / at risk) | 79/604 | 79/507
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=604) | Alternative TNFi (N=507)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 8 | 8
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 4 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 0
Abscess limb (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Genital infection female (Infections and infestations) | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina unstable (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Myopericarditis (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Sigmoiditis (Gastrointestinal disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest pain (General disorders) | 2 | 1
Device dislocation (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Quadriparesis (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 2 | 0
Abdominal hernia repair (Surgical and medical procedures) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0
Joint fluid drainage (Surgical and medical procedures) | 1 | 0
Urethral meatotomy (Surgical and medical procedures) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Depression (Psychiatric disorders) | 0 | 2
Completed suicide (Psychiatric disorders) | 0 | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=604) | Alternative TNFi (N=507)
Diarrhoea (Gastrointestinal disorders) | 5 | 12
Nausea (Gastrointestinal disorders) | 12 | 13
Lower respiratory tract infection (Infections and infestations) | 14 | 10
Urinary tract infection (Infections and infestations) | 25 | 16
Headache (Nervous system disorders) | 15 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Rash (Skin and subcutaneous tissue disorders) | 8 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.